CLINICAL TRIAL: NCT06826495
Title: Thiol Disulfide Balance and Oxidative Stress Change in Endometrial Polyp Patients
Status: Completed | Type: Observational
Sponsor: Mardin Artuklu University (Other)
Responsible Party: Principal Investigator, Hasan Basri Savas, Associate Professor, Mardin Artuklu University
Other Study IDs: 10354421-2020/23-8
Record Dates: First submitted 2025-02-07; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Endometrial Polyp; Oxidative Stress

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- endometrial polyps: Women with endometrial polyp
- control group: Participants in the control group were confirmed to be free of endometrial polyps via TVUSG and saline infusion ultrasonography

SUMMARY:
Changes in Thiol Disulfide Balance and Oxidative Stress Mechanisms in Patients with Endometrial Polyps

ELIGIBILITY:
Inclusion Criteria:

For participants in the control group:

• To be without endometrial polyp

For the polyp group, they were as follows:

* Individuals experiencing menometrorrhagia
* A body mass index (BMI) of 25 or more
* Hypertension
* Endometrial polyps detected via saline infusion ultrasonography

Exclusion Criteria:

* Pregnancy
* Diabetes mellitus
* Pelvic mass
* Malignancy
* The use of Tamoxifen, hormonal contraceptives, or hormone replacement therapy.

Ages: 20 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: A total of fifty-four participants, aged 20 to 48, took part in the study, including twenty-four women diagnosed with endometrial polyps and thirty women as the control group.
Sampling Method: Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2021-01-02 (Actual); Primary Completion 2022-01-03 (Actual); Study Completion 2022-01-05 (Actual)

PRIMARY OUTCOMES:
Oxidative stress markers | From January 2021 to January 2022
  Total antioxidant status (μmol Trolox equivalent/ L)
Oxidative stress markers | From January 2021 to January 2022
  Total oxidant status (μmol H2O2 equivalent/L)
Oxidative stress markers | From January 2021 to January 2022
  Oxidative stress index (arbitrary unit)
Oxidative stress markers | From January 2021 to January 2022
  Paraoxonase (U/L)
Oxidative stress markers | From January 2021 to January 2022
  Arylesterase (Ku/l)
Oxidative stress markers | From January 2021 to January 2022
  Total thiol (µmol / L)
Oxidative stress markers | From January 2021 to January 2022
  Native thiol (µmol / L) / alb (g / l)
Oxidative stress markers | From January 2021 to January 2022
  Disulfide (-S-S-) (µmol / L) / alb (g/l)
Oxidative stress markers | From January 2021 to January 2022
  Ischemia-modified albumin (u/L)

CONTACTS AND LOCATIONS:
Locations (1):
- Alanya Training and Research Hospital Gynecology and Obstetrics Department, Antalya, Turkey (Türkiye)